CLINICAL TRIAL: NCT05256862
Title: Improving Cervical Cancer Screening in Women Living With HIV Attending Chronic Disease Clinics in Semi-rural Tanzania
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Krebsforschung Schweiz, Bern, Switzerland (Other); Abviris Deutschland GmbH (Unknown); Charité-University Medicine (Berlin, Germany) (Unknown); Swiss Tropical and Public Health Institute (Switzerland) (Unknown)
Responsible Party: Sponsor
Other Study IDs: AO_2021-00006; bb22Kind
Record Dates: First submitted 2022-02-10; First posted 2022-02-25 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Cervical Cancer Screening
Keywords: women living with HIV (WLWH); cervical cancer; cervical cancer prevention clinic; cervical intraepithelial neoplasia; Human Papilloma Virus; Human Immunodeficiency Virus; Squamous Intraepithelial Lesion; Kilombero and Ulanga Anti-retroviral Cohort; QuantiGene-molecular profiling histology
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia; Acquired Immunodeficiency Syndrome; Squamous Intraepithelial Lesions | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection — Data collection
  * on the effect of a bundle of measures on the proportion of females being screened for cervical cancer in the Kilombero and Ulanga Antiretroviral Cohort (KIULARCO) comparing the time period before implementation (01/2017-01/2020) and after implementation (02/2020-06/2022)
  * on the performance of three novel tests as triage tool in the screening algorithm, QG-MPH, Prevo-check® and PT Monitor®

SUMMARY:
This study is to analyse the effect of a bundle of measures on the proportion of females being screened for cervical cancer in the Kilombero and Ulanga Antiretroviral Cohort (KIULARCO), comparing the time period before implementation (01/2017-01/2020) and after implementation (02/2020-06/2022). It is to assess the performance of two novel diagnostic tests (QuantiGene-molecular profiling histology (QG-MPH) and PT Monitor® immunoassay) and established tests (Seegene Anyplex™ II 28 HPV Test and Prevo-check®) as potential triage tests for the development of future clinical decision algorithms for CC screening.

DETAILED DESCRIPTION:
Cervical cancer (CC) is the most common cancer among women living with HIV (WLWH) and the leading cause of cancer-related death in women in East Africa. Currently there are around 2800 WLWH in care at the Chronic Disease Clinic of Ifakara (CDCI), of whom only 8% attended CC screening services in the last three years.

This research project is to assess (with a mixed-method, before-/after-study) the impact of a bundle of procedures, which consists of: portable colposcopy, Human Papilloma Virus (HPV) testing and treatment of precancerous cervical lesions by Loop electrosurgical excision procedure (LEEP).

This study is also to analyze the prevalence of cervical disease in the cohort, stratified by stage and co-infections, as well as the acceptability, feasibility and costs.

Additionally, it will assess the performance of two novel diagnostic tests (QG-MPH and PT Monitor® immunoassay) and established tests (Seegene Anyplex™ II 28 HPV Test and Prevo-check®) as potential triage tests for the development of future clinical decision algorithms for CC screening. This is an implementational study nested within the KIULARCO study consisting of two interacting parts: a pre/post assessment of the impact of the bundle of interventions with mixed-methods study design and the diagnostic tests accuracy (evaluated with a cross-sectional study). The treatment investigated is regarded as standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* WLWH enrolled in KIULARCO, who are at least 3 months on Anti-Retroviral Treatment (ART)
* 18-65 years of age
* Non-pregnant (reported)
* Signed informed consent

Exclusion Criteria:

* Pregnancy
* Known invasive cervical cancer
* Any condition interfering with visualization of the cervix

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women will be informed during their routine control within HIV care about the study on improved CC screening procedures and referred to the study team if consenting.
  All interventions will be offered routinely to patients, but are not mandatory if they refuse them. Patients not consenting will be advised to seek regular services for CC screening according to the national guidelines. Apart from routine clinical visits, no additional visits are scheduled for this study unless medically indicated.
Sampling Method: Probability Sample
Enrollment: 2974 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-10-18 (Actual)

PRIMARY OUTCOMES:
Number of WLWH attending CC screening | one time assessment at Screening
  Number of WLWH attending CC screening in the period 08/2021 - 06/2022; Attendance of screening: for the pre-phase women undergoing Visual inspection with acetic acid (VIA), for the post- phase women performing cervical self-sampling.

SECONDARY OUTCOMES:
Number of detected High Grade Squamous Intraepithelial Lesion /Cervical Cancer (HSIL/CC) in cervical self-samples by QuantiGene-molecular profiling histology (QG-MPH) | one time assessment at Screening
  Diagnostic test accuracy in detecting High Grade Squamous Intraepithelial Lesion /Cervical Cancer (HSIL/CC) in cervical self-samples by QuantiGene-molecular profiling histology (QG-MPH)
Number of detected patients with Human Papilloma Virus (HPV) 16 and 18 induced Cervical Intraepithelial Neoplasia grade 3 or above (CIN3+) by Serum PT Monitor®. | one time assessment at Screening
  Diagnostic test accuracy in detecting patients with Human Papilloma Virus (HPV) 16 and 18 induced Cervical Intraepithelial Neoplasia grade 3 or above (CIN3+) by Serum PT Monitor®.

CONTACTS AND LOCATIONS:
Overall Officials: Ivana Di Salvo, MD, Principal Investigator — University Women's Hospital Basel
Locations (1):
- Saint Francis Referral Hospital, Ifakara Health Institute (IHI, United Republic of Tanzania), Ifakara, Tanzania

REFERENCES:
- [Derived] Di Salvo I, Mnzava D, Nicoletti GJ, Senkoro E, Ndege RC, Huang DJ, Makunja NT, Kassiga GI, Kaufmann AM, Weisser M, Kind AB. Upscaling cervical cancer screening and treatment for women living with HIV at a rural referral hospital in Tanzania: protocol of a before-and-after study exploring HPV testing and novel diagnostics. BMC Health Serv Res. 2023 Mar 10;23(1):234. doi: 10.1186/s12913-023-09113-3. PMID 36894985